CLINICAL TRIAL: NCT04241276
Title: Phase IIb Randomised Clinical Trial Repurposing ATRA as a Stromal Targeting Agent in a Novel Drug Combination for Pancreatic Cancer
Brief Title: A Randomised Trial of ATRA in a Novel Drug Combination for Pancreatic Cancer
Acronym: STARPAC2
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Medical Research Council (Other Government); Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 274948
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Tretinoin; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gemcitabine + nab-paclitaxel (Active Comparator): Patients will receive Gemcitabine and nab-Paclitaxel in 28 day cycles until disease progression.
  Interventions: Drug: Gemcitabine; Drug: nab-paclitaxel
- Gemcitabine + nab-paclitaxel + ATRA (Experimental): Patients will receive ATRA, Gemcitabine and nab-Paclitaxel in 28 day cycles. ATRA will be administered for 6 cycles whereas Gemcitabine/nab-Paclitaxel will be administered until disease progression.
  Interventions: Drug: ATRA; Drug: Gemcitabine; Drug: nab-paclitaxel

INTERVENTIONS:
Drug: ATRA — 45 mg/m2 orally (in two divided doses) from days 1 to 15 of each cycle
  Other Names: Tretinoin; Vesanoid
  Arms: Gemcitabine + nab-paclitaxel + ATRA
Drug: Gemcitabine — 1000mg/m2 IV on days 1, 8 and 15 of a 28 day cycle
Drug: nab-paclitaxel — 125mg/m2 IV on days 1, 8 and 15 of a 28 day cycle
  Other Names: Abraxane

SUMMARY:
This is an open-label, multi-centre, randomised, stratified, phase IIb clinical trial of ATRA administered in combination with gemcitabine and nab-paclitaxel in patients with laPDAC.

DETAILED DESCRIPTION:
Patients will be randomised to receive gemcitabine + nab-paclitaxel or gemcitabine + nab-paclitaxel + ATRA. Treatment will be administered in 28 day cycles. ATRA will be administered for 6 cycles whereas gemcitabine/nab-paclitaxel will be administered until disease progression. Treatment may be discontinued earlier due to unacceptable toxicities or death or because the patient requests to be withdrawn from study treatment. If treatment with gemcitabine/nab-paclitaxel is stopped prior to the patient completing 6 cycles of treatment with ATRA (if allocated), the patient may continue on treatment with ATRA alone until the 6 cycles are completed, at the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following inclusion criteria to be enrolled in the study:

1. Written informed consent prior to admission to this study
2. Age ≥16 years. No upper age limit.
3. ECOG performance status 0 or 1
4. Histologically proven pancreatic ductal adenocarcinoma (PDAC) as part of the Precision-Panc Master Protocol, or for patients who have gone exploratory laparotomy and found to have locally, unresectable advanced disease.
5. Locally advanced disease which is measurable according to the Response Evaluation Criteria in Solid Tumours (RECIST v1.1).
6. CT chest abdomen and pelvis as well as PET-CT within 28 days of day 1 of treatment (MRI Liver only if indeterminate liver lesions) to confirm absence of metastatic disease.
7. Received no prior systemic therapy for pancreatic cancer.
8. Adequate haematologic and end organ function, defined by the following laboratory results obtained within 14 days prior to the first study treatment:

   1. Absolute Neutrophil Count ≥ 1.5 x 109/l (without granulocyte colony-stimulating factor support within 2 weeks prior to the first study treatment)
   2. Platelet count ≥ 100 x 109/l (without transfusion within 2 weeks prior to the first study treatment)
   3. Haemoglobin ≥ 10 g/dl (transfusion permitted to establish target haemoglobin levels prior to the first study treatment)
   4. Calculated creatinine clearance (e.g. Cockcroft-Gault) ≥ 50 ml/min
   5. Bilirubin level ≤ 1.5 ULN (patients with known Gilbert disease who have bilirubin levels ≤ 3 x ULN may be enrolled). Patients must be able to undergo biliary stenting if required before or, if required, during the trial
   6. AST or ALT <2.5 x ULN
   7. Alkaline phosphatase (ALP) <2.5 x ULN
   8. INR and aPTT ≤1.5 x ULN; this applies only to patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose.
9. Female patients of child-bearing potential are eligible, provided they have a negative serum pregnancy test within 7 days prior to the first dose of study treatment, preferably as close to the first dose as possible. All patients with reproductive potential must agree to use a medically acceptable method of contraception throughout the treatment period and for 1 month after discontinuation of ATRA and / or gemcitabine/nab-paclitaxel (whichever is the latest) and for 6 months after discontinuation for male patients. Acceptable methods of contraception include IUD, oral contraceptive, sub-dermal implant and double barrier (condom with a contraceptive sponge or contraceptive pessary). Micro-dosed progesterone preparations ("mini-pill") are an inadequate method of contraception during treatment with ATRA. If patients are taking this pill they should be instructed to stop and another form of contraceptive should be prescribed instead.
10. Able to follow protocol requirements as assessed by the Principal Investigator.

Exclusion Criteria:

A patient will not be eligible for inclusion in this study if any of the following criteria apply:

1. Patient has known distant metastases.
2. Patient has experienced a significant reduction in performance status between the screening/ baseline visit and within 72 hours prior to commencement of treatment as per trial protocol, such that the ECOG PS is ≥ 2 as per the Investigator's assessment.
3. Patients with pre-existing sensory neuropathy >grade 1
4. History of other malignancies (except cured basal or squamous cell carcinoma, superficial bladder cancer, prostate cancer in active surveillance, or carcinoma in situ of the cervix) unless documented free of cancer for ≥2 years
5. Patient has active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy.
6. Patient has known active, uncontrolled HIV, or active, uncontrolled hepatitis B or C infection. Patients with undetectable viral load are eligible.
7. Patient has undergone major surgery, other than diagnostic surgery (i.e., surgery done to obtain a biopsy for diagnosis without removal of an organ), within 4 weeks prior to Day 1 of treatment in this study.
8. Patient has a history of allergy (including soya bean or peanut allergies) or hypersensitivity to any of the study drugs or any of their excipients, or the patient exhibits any of the events outlined in the Contraindications or Special Warnings and Precautions sections of the products or comparator SmPC or Prescribing Information.
9. History of connective tissue disorders (e.g., lupus, scleroderma, arteritis nodosa).
10. Patient with a history of interstitial lung disease, history of slowly progressive dyspnoea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis or multiple allergies.
11. Patient with high cardiovascular risk , including, but not limited to, recent coronary stenting or myocardial infarction in the past year.
12. History of Peripheral Artery Disease (e.g., claudication, Leo-Buerger's disease).
13. Patient has serious medical risk factors involving any of the major organ systems, or serious psychiatric disorders, which could compromise the patient's safety or the study data integrity.
14. Concurrent treatment with other experimental drugs or participation in another clinical trial with any investigational drug at least ≤30 days prior to study entry depending on the half-life of the investigational drug and/or guidance issued by the IMP manufacturer.
15. Patient is taking any prohibited concurrent medication, including vitamin A supplements, and is unwilling to stop use prior to and during the trial.
16. Patient is pregnant, planning to become pregnant or breast feeding.
17. Patient has received a live vaccine within four weeks prior to receiving their first dose of study treatment.
18. Patient is unwilling or unable to comply with study procedures, as assessed by the Principal Investigator.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2020-04-30 (Actual); Primary Completion 2028-06-29 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy of ATRA when given in combination with gemcitabine and nab-paclitaxel based on progression free survival (PFS). | Assessed 8 weekly until progression or death or end of trial, whichever comes first
  PFS defined as the time from the date of randomisation to the date of first documented tumour progression or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
To assess the efficacy of ATRA when given in combination with gemcitabine and nab-paclitaxel based on objective response rate (ORR). | Assessed 8 weekly until progression or death or end of trial, whichever comes first
  ORR defined as the number of patients with an objective response (OR) divided by the number of patients analysed. OR is defined as the number of patients with at least one confirmed response of complete response (CR) or partial response (PR). OR will be calculated in patients with measurable disease at baseline.
To assess the efficacy of ATRA when given in combination with gemcitabine and nab-paclitaxel based on overall survival (OS). | Assessed 8 weekly until progression or death and then 3 monthly for at least 12 months after the last safety visit
  OS is defined as the time from the date of randomisation to death from any cause.
To assess the safety and tolerability of ATRA when given in combination with gemcitabine and nab-paclitaxel over the first 6 cycles. | 6 cycles (1 cycle = 28 days)
  The worst recorded toxicity grade for each patient on the NCI-CTCAE toxicity scale (version 5.0) over the first 6 cycles of treatment
To assess the surgical resection rate of ATRA when given in combination with gemcitabine and nab-paclitaxel. | From consent to at least 12 months after the last safety visit, but further if required as per physician decision - through study completion
  Surgical resection rate defined as patients undergoing complete resection of known pancreatic primary and associated lymph nodes at any point after enrolment, in each arm.
To assess the resection margin negative (R0) surgical resection rate of ATRA when given in combination with gemcitabine and nab-paclitaxel. | From consent to at least 12 months after the last safety visit, but further if required as per physician decision - through study completion
  R0 surgical resection rate defined as histologically confirmed complete resection of known pancreatic primary from those resected.
To assess quality of life (QOL) of patients receiving ATRA in combination with Gemcitabine and Nab-Paclitaxel: EQ-5D-5L | Assessed at the beginning of each cycle until progression (1 cycle = 28 days)
  QoL scores for the five dimensions of the EQ-5D-5L (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) will be used to calculate weighted health status scores.

CONTACTS AND LOCATIONS:
Overall Officials: Hemant Kocher, Professor, Study Chair — Queen Mary University of London
Locations (1):
- Barts NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kocher HM; BCI-STARPAC2 team; BPTB team; Precision-Panc team; Sasieni P, Corrie P, McNamara MG, Sarker D, Froeling FEM, Christie A, Gillmore R, Khan K, Propper D. Study protocol: multi-centre, randomised controlled clinical trial exploring stromal targeting in locally advanced pancreatic cancer; STARPAC2. BMC Cancer. 2025 Jan 20;25(1):106. doi: 10.1186/s12885-024-13333-z. PMID 39833722